CLINICAL TRIAL: NCT03618446
Title: Predictors Of Mortality After Pelvic Fractures: A Retrospective Cohort Study From A Level-1 Trauma Center In Upper Egypt.
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Collaborators: AO Clinical Investigation and Publishing Documentation (Other)
Responsible Party: Principal Investigator, Osama Farouk, Professor of Orthopaedic and Trauma Surgery, Assiut University
Other Study IDs: 17100526
Record Dates: First submitted 2018-07-05; First posted 2018-08-07 (Actual); Last update posted 2022-02-16 (Actual); Status verified 2022-02

CONDITIONS: Registries; Pelvic Bone Injury; Morality
Keywords: Pelvic fractures; mortality; predictors; trauma registry
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Survivors: Patients whose pelvic fracture and survived till time of discharge from the hospital.
  Interventions: Other: The presence of a pelvic fracture
- Non-Survivors: Patients whose pelvic fracture and died while in hospital.
  Interventions: Other: The presence of a pelvic fracture

INTERVENTIONS:
Other: The presence of a pelvic fracture

SUMMARY:
A retrospective cohort study was carried out for all pelvic fracture patients admitted to Assiut University Trauma Unit (AUTU), a level-1 trauma center. (AUTU) is located in Upper Egypt and provides healthcare to over 30,000 patients per year.

DETAILED DESCRIPTION:
In 2010, a Pelvic Injury Registry was developed to document treatment and outcomes in a standardized manner. All patients admitted to AUTU sign an informed consent to permit using their data for research purposes. Patients' data are prospectively collected and stored in a local database specifically designed for this purpose.

Data collected included age, gender, mechanism of injury, fracture classification, associated injuries, and admission to ICU, the length of hospital stay and presence of abdominopelvic collection as diagnosed by Focused Assessment with Sonography for Trauma (FAST) at admission. The primary outcome measure was in-hospital mortality. Predictors of in-hospital mortality were identified by comparing characters of survivors and non-survivors. Secondary objectives were to analyse the differences between adults and children and to analyse the causes and timing of death.

ELIGIBILITY:
Inclusion Criteria:

* first-time admissions and patients whose treatment was completed at our hospital
* all pelvic fracture patients admitted to our Trauma Unit.

Exclusion Criteria:

* penetrating injuries
* isolated acetabular fractures
* Patients who were discharged on their own will against the medical advice or whose treatment was continued at another hospital
* re-admitted patients
* Firearm injuries

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: 1188 patients were considered eligible for analysis. These were further divided into an adult cohort whose age is above 16 years (951 patients) and a pediatric cohort (237 patients).
Sampling Method: Probability Sample
Enrollment: 1188 (Actual)
Dates: Start 2010-01-01 (Actual); Primary Completion 2013-12-31 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
in-hospital mortality | One month
  Death occurring while the patient is admitted in the hospital.

CONTACTS AND LOCATIONS:
Overall Officials: Osama Farouk, Principal Investigator — Assiut University